CLINICAL TRIAL: NCT06601699
Title: Neuromodulation-assisted Ego-disengagement: The NEURO-EGO Study
Brief Title: Neuromodulation-assisted Ego-disengagement: The NEURO-EGO Study Stage 2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Tiny Blue Dot Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: 2023-0613 Stage 2; A535100 (Other: UW Madison); Protocol Version 10/9/2025 (Other: UW Madison)
Record Dates: First submitted 2024-09-10; First posted 2024-09-19 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Healthy
Keywords: meditation; brain stimulation
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Stimulation (Experimental): Participants will undergo TES or TES-TI stimulation in 5-minute blocks up to eight times a day on three separate days each separated by one week.
  Interventions: Device: Transcranial electrical stimulation (TES); Device: Transcranial electrical stimulation with temporal interference (TES-TI)
- Sham stimulation (Sham Comparator): Participants will undergo sham stimulation in 5-minute blocks up to eight times a day on three separate days each separated by one week.
  Interventions: Device: Transcranial electrical stimulation (TES); Device: Transcranial electrical stimulation with temporal interference (TES-TI)

INTERVENTIONS:
Device: Transcranial electrical stimulation (TES) — TES uses specific electrode arrangement patterns to selectively stimulate the brain. Participants will wear an hdEEG (high density electroencephalography) cap which will allow intermittent periods of stimulation from TES.
Device: Transcranial electrical stimulation with temporal interference (TES-TI) — TES-TI uses specific electrode arrangement patterns to selectively stimulate the brain. Participants will wear an hdEEG (high density electroencephalography) cap which will allow intermittent periods of stimulation from TES-TI.

SUMMARY:
The goal of this clinical trial is to learn whether brain stimulation technology can help people reach a meditative state quickly and easily without years of meditation training. The researchers want to see if this will help people distance themselves from their thoughts and feeling, and if this will lead to improvements in openness and wellbeing the same way meditation can.

Participants will:

* Complete questionnaires
* Perform a guided meditation task (The Bell Task)
* Wear a high density electrocochleography (hdEEG) cap
* Undergo brain stimulation

DETAILED DESCRIPTION:
This study is being done to evaluate the relative effectiveness of distinct types of non-invasive brain stimulation - NIBS (TES-TI and TES) on subjective ego disengagement and cortical activity in experienced meditators and meditation naïve healthy adults.

Stage 1a was designed to establish the optimal level of stimulation to achieve ego displacement in experienced meditators. Stage 1b used the level of stimulation established in 1a to discern the region of the posteromedial cortex (PMC) where disruption is most effective in achieving ego displacement in experienced meditators. This stage, stage 2 will use the most effective stimulation and PMC parameters to meditation naïve healthy adults.

Primary Objective (stage 2):

- To evaluate the effectiveness of NIBS on ego disengagement and cortical activity in meditation naïve healthy adults acutely and longitudinally

Secondary Objectives (stage 2):

* Evaluate the relationships between NIBS, ego-disengagement, and trait assessments openness and wellbeing
* Evaluate the effect of the use of topical anesthetics on the EEG response evoked by NIBS

ELIGIBILITY:
Inclusion Criteria:

* Adults, ages 18 to 80 of any identified gender
* Medically healthy
* English-speaking (able to provide consent and complete questionnaires)
* Healthy adults who are meditation-naïve
* Citizen or legal resident

Exclusion Criteria:

* Any current or past history of neurological disorders or acquired neurological disease (e.g. stroke, traumatic brain injury), including intracranial lesions
* Any current or past history of bipolar disorder and/or hypomania
* Any current or past history of psychosis
* History of head trauma resulting in prolonged loss of consciousness; or a history of great than 3 grade I concussions
* Current history of poorly controlled headaches including intractable or poorly controlled migraines
* Any systemic illness or unstable medical condition that may cause a medical emergency in case of a provoked seizure (cardiac malformation, cardiac dysrhythmia, asthma, etc.)
* History of fainting spells of unknown or undetermined etiology that might constitute seizures
* History of seizures, diagnosis of epilepsy, history of abnormal (epileptiform) EEG, or family history of treatment resistant epilepsy with the exception of a single seizure of benign etiology (e.g. febrile seizures) in the judgment of a board-certified neurologist
* Possible pregnancy. All female participants of child-bearing age are required to have a pregnancy test
* Any metal in the brain, skull or head
* Any contraindications to MRI
* Any medical devices or implants (i.e. cardiac pacemaker, medication infusion pump, cochlear implant, vagal nerve stimulator, dental implants (this includes a permanent retainer)) unless otherwise approved by the responsible MD
* Substance abuse or dependence within the past six months
* Any medication that may alter seizure threshold i.e., ADHD stimulants (Adderall, amphetamine); Tricyclic/atypical antidepressants (Amitriptyline, Dioxepine, Imipramine Maprotiline, Nortriptyline, Bupropion); Antipsychotics (Chlorpromazine, Clozapine), Bronchodilators (theophylline, aminophylline); Antibiotics (fluoroquinolones, imipenem, penicillin, cephalosporins, metronidazole, isoniazid); Antiviral (Valacyclovir, Ritonavir); OTC (Diphenhydramine)
* Claustrophobia (a fear of small or closed places)
* Back problems that would prevent lying flat for up to two hours
* Having experienced a traumatic event that caused lasting distress or required treatment
* Motion sickness
* Any hair braid, dreadlocks, hair pieces, or extensions which cannot be taken out or adjusted to permit comfortable and comprehensive participation before the MRI scans and/or stimulation sessions
* Any head coverings or headdress that participant feels uncomfortable removing for the purposes of the MRI scans and/or stimulation session

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-08-27 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Ego-Disengagement scale | baseline, week 1, week 2, week 3, week 7
  Ego-disengagement will be measured using the bell task. This meditation task consists of five "bell trials." During each trial, subjects will be asked to focus on the sound of a bell until it fades, then on the space left empty by the faded sound, resting free from thoughts as long as possible (meditation condition). Afterward, subjects will respond to a few questions designed to assess their level of ego-disengagement during the trials. This is a five-question form that asks subjects to rate, on a scale from 0-4, the degree to which they were perceiving something, imagining something, thinking about themselves, or thinking about something during the previous bell trial and then to rate the valence of their emotional state during the trial from 1 (highly negative) to 6 (highly positive).
Cortical activity - change in gamma band power | week 1, week 2, week 3, final visit (week 7)
  Gamma band power will be measured with hdEEG during stimulation. A decrease indicates greater level of ego disengagement.

SECONDARY OUTCOMES:
Change in Big Five Aspects Scale (BFAS) | baseline to week 3
  This is a 44-item inventory that measures five different personality traits by asking subjects to respond to various items (e.g., I see myself as someone who is talkative) on a scale from 1 (disagree strongly) to 5 (agree strongly).
Change in Fulfilled Life Scale (FLS) | baseline to week 3
  This is a 32-item inventory that asks subjects to respond to various items (e.g., When I look back on my life, I feel deep inner contentment) on a scale from 1 (does not apply at all) to 6 (applies completely) and is designed to assess subjects' feelings of having lived a full life.
Change in PROMIS Anxiety | baseline to week 3
  This is an 8-item inventory asking subjects to rate from 1-5 the frequency with which they have experienced components of anxiety in the last seven days. Higher scores reflect greater anxiety.
Change in PROMIS Depression | baseline to week 3
  This is an 8-item inventory asking subjects to rate from 1-5 the frequency with which they have experienced components of depression in the last seven days. Higher scores reflect greater depression.
Change in Perceived Stress Scale (PSS) | baseline to week 3
  This is a 10-item inventory asking subjects to rate from 0-4 the frequency with which they have felt various kinds of stress in the last month. Participants rate each item on a scale ranging from Never (0) to Very often (4). Seven of the items with positive statements are scored in reverse. As the scores obtained from the scale increase, the perceived stress level of the person increases. Scores range from 0-40.
Change in Questionnaire for Eudaimonic Well-Being (QEWB) | baseline to week 3
  This is a 21-item inventory asking subjects to rate from 0-4 the extent to which they agree with various statements designed to assess their overall well-being. Scores range from 0-84 with higher scores indicating higher levels of well-being.
Cortical activity - change in alpha band power (topical anesthetic vs. no topical anesthetic) | week 1, week 2, week 3, final visit (week 7)
  Alpha band power will be measured with hdEEG during stimulation. An increase indicates greater level of ego disengagement. Cortical activity will be compared between sessions that use topical anesthetics and those that do not use topical anesthetics below the sensors to evaluate whether skin receptors are a confounding factor.
Cortical activity - change in gamma band power (topical anesthetic vs. no topical anesthetic) | week 1, week 2, week 3, final visit (week 7)
  Gamma band power will be measured with hdEEG during stimulation. A decrease indicates greater level of ego disengagement. Cortical activity will be compared between sessions that use topical anesthetics and those that do not use topical anesthetics below the sensors to evaluate whether skin receptors are a confounding factor.

CONTACTS AND LOCATIONS:
Overall Officials: Melanie Boly, MD, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No